CLINICAL TRIAL: NCT07127913
Title: Closed-Loop Deep Brain Stimulation for Bipolar Depression (PReSiDio-BP)
Brief Title: Closed-Loop Deep Brain Stimulation for Treatment-Resistant Bipolar Depression
Acronym: PReSiDio-BP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Andrew Krystal (Other)
Responsible Party: Sponsor-Investigator, Andrew Krystal, Professor of Psychiatry and Behavioral Sciences, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 17-23724B
Record Dates: First submitted 2025-08-01; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Bipolar II Disorder; Bipolar II Disorder, Most Recent Episode Major Depressive
Keywords: Bipolar II Disorder; Depression; Treatment-resistance; Deep brain stimulation; Closed-loop; Biomarker; Responsive neurostimulation; Brain surgery
MeSH Terms: conditions — Bipolar Disorder; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Experimental: Arm 1: Intervention (stimulation ON) (Experimental): This is a crossover trial. Each patient will receive 12 wks of stimulation ON (arm 1), stimulation OFF (arm 2), and Stimulation ON Active Control (fixed intermittent) (arm 3) in random order.
  Interventions: Device: Device: Stimulation-ON
- Sham Comparator: Arm 2: Sham Control (stimulation OFF) (Sham Comparator): This is a crossover trial. Each patient will receive 12 wks of stimulation ON (arm 1), stimulation OFF (arm 2), and Stimulation ON Active Control (fixed intermittent) (arm 3) in random order.
  Interventions: Device: Device: Stimulation-OFF
- Active Comparator: Arm 3: Active Control (stimulation ON fixed intermittent) (Active Comparator): This is a crossover trial. Each patient will receive 12 wks of stimulation ON (arm 1), stimulation OFF (arm 2), and Stimulation ON Active Control (fixed intermittent) (arm 3) in random order.
  Interventions: Device: Device: Stimulation -ON Active Control

INTERVENTIONS:
Device: Device: Stimulation-ON — Active neurostimulation from the NeuroPace RNS® System triggered by a biomarker
  Arms: Experimental: Arm 1: Intervention (stimulation ON)
Device: Device: Stimulation-OFF — No neurostimulation from the NeuroPace RNS® System
  Arms: Sham Comparator: Arm 2: Sham Control (stimulation OFF)
Device: Device: Stimulation -ON Active Control — Active neurostimulation from the NeuroPace RNS® System triggered with a fixed duty cycle
  Arms: Active Comparator: Arm 3: Active Control (stimulation ON fixed intermittent)

SUMMARY:
Neurons are specialized types of cells that are responsible for carrying out the functions of the brain. Neurons communicate with electrical signals. In diseases such as major depression this electrical communication can go awry. One way to change brain function is using electrical stimulation to help alter the communication between groups of neurons in the brain.

The purpose of this study is to test a personalized approach to brain stimulation as an intervention for bipolar depression The study researchers will use a surgically implanted device to measure each individual's brain activity related to his/her depression. The researchers will then use small electrical impulses to alter that brain activity and measure whether these changes help reduce depression symptoms. This study is intended for patients with major depression whose symptoms have not been adequately treated with currently available therapies.

The device used in this study is called the NeuroPace Responsive Neurostimulation (RNS) System. It is currently FDA approved to treat patients with epilepsy. The study will test whether personalized responsive neurostimulation can safely and effectively treat bipolar depression.

DETAILED DESCRIPTION:
This is a single-center 3-stage feasibility study of personalized closed-loop stimulation for treatment resistant Bipolar Depression. Depending on participant's results at each stage, he/she might not be eligible to proceed to all 3 stages.

Stage 1 of the study will involve surgically implanting small, thin electrodes in brain regions that regulate depression in order to identify personalized treatment sites. The researchers will test stimulation in the different brain regions and their effect on bipolar depression symptoms. The electrodes will be surgically removed at the end of Stage 1.

Stage 2 will involve a second brain surgery to implant the NeuroPace RNS® System. Researchers will use information from Stage 1 to decide where to implant the electrodes of the RNS System. Over the next ~4-18 months, participants will have regular study visits in the clinic where the researchers will determine a personalized brain activity pattern that correlates with depression symptoms and can be paired with stimulation to improve depression symptoms.

Stage 3 will be 36-40 weeks long and will involve turning ON and OFF the intervention to test its effectiveness. Participants will have a variable start time for Stage 3 to facilitate blinding of both patients and clinician raters. This variable time will be randomized from conditions of 0 days, 2 weeks, or 4 weeks (during which time participants will remain on optimized closed-loop stimulation). Each participant will have three 12-week periods: closed-loop stimulation (intervention), open-loop/fixed intermittent stimulation (active control), and sham (passive control), order counterbalanced.

At the end of this stage the participant can choose to continue with long-term follow-up or have the RNS System surgically removed.

ELIGIBILITY:
Inclusion Criteria:

* Age 22-70
* Meet Diagnostic and Statistical Manual-V (DSM-V) diagnostic criteria for Bipolar II Disorder, with an episode of depression lasting at least 1 year that is treatment resistant as defined above, without a manic or hypomanic episode in the last 2 years; patients must be taking a mood stabilizer (lithium >0.6 mEq/L or valproate >350 mM/L), an atypical antipsychotic, or a combination of a mood stabilizer and an atypical antipsychotic for at least 2 weeks at a stable dosage before starting the study and must continue taking anti-manic medication throughout their participation in the study unless discontinuation is necessary because of patient safety/health considerations.
* Must have either failed ECT (it was effective but not tolerated due to side effects; it was effective, but patients could not achieve a sustained response), not been able to complete a course of ECT due to side effects, or have been medically advised to receive ECT and have been unwilling or unable to obtain ECT.
* Has MADRS score of > 26 at two baseline visits
* Ability to complete repeated administrations of MDD rating scales.
* If patient is on a regimen of psychotropic medication, no changes in this regimen should be expected during the 4 weeks prior to entry into and the duration of the study.
* Willing and able to undergo invasive brain recording/stimulation study
* Willing and able to attend multiple research visits and perform at-home research protocol
* Willing and able to provide informed consent
* Ability to speak and read English

Exclusion Criteria:

* Meets DSM-V criteria for a psychotic disorder, eating disorder, panic disorder, posttraumatic stress disorder, obsessive compulsive disorder, tic disorder, or another comorbid psychiatric disorder other than MDD or generalized anxiety disorder based on a SCID
* Generalized anxiety disorder is the primary DSM-V disorder during the current MDD episode
* Active suicidal ideation with intent and plan as defined by a score of 5 on the Columbia-Suicide Severity Rating Scale (C-SSRS)
* History of suicide attempt requiring hospitalization in previous 2 years.
* Meets criteria for alcohol or substance abuse or dependence (other than caffeine) in previous 6 months, determined by the SCID
* Has a personality disorder based on the investigator's assessment that the investigator believes will adversely impact subject compliance or safety
* Fibromyalgia or chronic fatigue syndrome
* Current condition requiring chronic narcotic use
* History of traumatic brain injury, another neurological disorder, or developmental delay
* History of seizures
* MRI (done within one year of the first visit) with significant abnormalities
* Previous ablative intracranial surgery or previously implanted deep brain stimulation system or any previously implanted device treatment involving brain stimulation
* Implantable hardware not compatible with MRI or with the study
* Major medical co-morbidities increasing the risk of surgery including severe diabetes, major organ system failure, history of hemorrhagic stroke, need for chronic anticoagulation other than aspirin, active infection, intracranial space occupying lesion, increased intracranial pressure, cardiovascular accident within the last month, aneurysm/abnormality, retinal detachment, unstable cardiovascular disease (recent myocardial infarction, severe ischemia, severe or uncontrolled hypertension), immunocompromised state, or malignancy with < 5 years life expectancy
* Inability to stop Coumadin or platelet anti-aggregation therapy for surgery and after surgery. - Patients taking these medications will need to discuss the need/risk of continuing these medications with their physicians and the PI or study personnel may contact the treating physician(s) to discuss the risks of anticoagulation/antiaggregation therapy discontinuation
* Coagulopathy. Patients will be excluded unless assessed and cleared by hematology
* Allergies or known hypersensitivity to materials in the NeuroPace RNS® System (i.e. titanium, polyurethane, silicone, polyetherimide, stainless steel)
* Subject lives alone without possibility of caregiver support post-hospital stay
* Inability to comply with study follow-up visits

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-07-16 (Actual); Primary Completion 2030-06-28 (Estimated); Study Completion 2035-06-28 (Estimated)

PRIMARY OUTCOMES:
Change in Montgomery-Asberg Depression Rating Scale (MADRS) score | Administered twice at baseline and every 2 weeks for the 36-40 weeks of Stage 3
  Effect size comparing closed-loop stimulation, open-loop (fixed intermittent) stimulation, and sham stimulation (MADRS score before and after each treatment period of the crossover). Higher MADRS score indicates more severe depression; the overall score ranges from 0 to 60.

SECONDARY OUTCOMES:
Change in Hamilton Depression Rating Scale (HAMD-17) score | Administered at baseline and every 4 weeks for the 36-40 weeks of Stage 3
  Effect size comparing closed-loop stimulation, open-loop (fixed intermittent) stimulation, and sham stimulation (HAMD-17 score before and after each treatment period of the crossover). The score for Hamilton Depression Rating Scale ranges from 0-50, with a higher score indicating more severe depression.
Change in the Inventory of Depressive Symptomatology Self-Report (IDS-SR) score | Administered at baseline and every 4 weeks for the 36-40 weeks of Stage 3
  Effect size comparing closed-loop stimulation, open-loop (fixed intermittent) stimulation, and sham stimulation (IDS-SR score before and after each treatment period of the crossover). The scores range from 0 to 27, with higher scores indicating more depressive symptoms.

OTHER OUTCOMES:
Daily stimulation events | Up to 24 weeks
  Number of daily stimulation events
Stimulation duration | Up to 24 weeks
  Cumulative stimulation duration per day
Stimulation site identification | Decision made in the 1-3 months following Stage 1
  The number of patients that move from Stage 1 to Stage 2 (stimulation site identified that acutely improved symptoms)
Biomarker identification in Stage 1 | Decision made in the 1-3 months following Stage 1
  Number of patients in whom we can identify a neural biomarker
Number of patients who had viable biomarker(s) identified in Stage 2 | Once at the end of Stage 2, ranging from 4-15 months
  Number of patients in whom we can utilize the biomarker to drive stimulation events using the RNS® System
Number and severity of adverse events | Through study completion, average of 2.5-3 years
  The number and type of serious adverse events that occur in comparison to comparable deep brain stimulation trials

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Krystal, MD, MS, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No